CLINICAL TRIAL: NCT03089606
Title: Pembrolizumab in Systemic Treatment-Naïve Distant Metastatic Melanoma and Exploration of Use of Baseline 11C-methyl-L-tryptophan (C11-AMT) PET Imaging as a Predictive Imaging Biomarker of Antitumor Response
Brief Title: Pembrolizumab TX-naive Distant Mets Melanoma and Use of (C11-AMT) PET at Baseline as Imaging Biomarker
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LCCC 1531
Record Dates: First submitted 2017-02-24; First posted 2017-03-24 (Actual); Results first posted 2022-07-14 (Actual); Last update posted 2023-11-15 (Actual); Status verified 2023-11

CONDITIONS: Melanoma
MeSH Terms: conditions — Melanoma | interventions — pembrolizumab; Tomography, X-Ray Computed

STUDY DESIGN:
Intervention Model Description: This is a phase 2, single-arm, open-label study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Single Arm (Other): This is a single arm study. All participants completed the study interventions which are pembrolizumab treatment, FDG PET, C11-AMT PET and CT scans.
  Interventions: Diagnostic Test: FDG PET/CT scan; Diagnostic Test: C11-AMT PET scan; Drug: Pembrolizumab; Diagnostic Test: CT scan

INTERVENTIONS:
Diagnostic Test: FDG PET/CT scan — 18F-fluorodeoxy glucose (FDG) positron emission tomography (PET) with intravenous (IV) contrast images are obtained before and at the end study treatment (pembrolizumab infusion).
Diagnostic Test: C11-AMT PET scan — 11C-methyl-L-tryptophan (C11-AMT) positron emission tomography (PET) images are obtained before study treatment (pembrolizumab infusion).
Drug: Pembrolizumab — 200 mg Pembrolizumab IV administered over 30 minutes on day 1. Repeat every 3 weeks for 4 cycles, until progression, or subject withdrawal for other reasons
  Other Names: Keytruda
Diagnostic Test: CT scan — Computerized tomography (CT) images are taken without IV contrast before the treatment (pembrolizumab infusion) and with IV contrast 3 months after the treatment start.

SUMMARY:
Explore the association between intensity of 11C-methyl-L-tryptophan (C11-AMT) positron emission tomography (PET) at baseline, as measured by mean standardized uptake value (SUVmax) at each lesion, total tumor metabolic volume, measurement of intra-tumoral and inter-lesional heterogeneity, with objective response rate (ORR) at 12 weeks (as defined via RECIST 1.1) to pembrolizumab in patients with treatment-naïve metastatic melanoma.

DETAILED DESCRIPTION:
Objectives:

Primary Objective

Explore the association between intensity of C11-AMT PET at baseline, as measured by mean standardized uptake value (SUVmax at each lesion), total tumor metabolic volume, measurement of intra-tumoral and inter-lesional heterogeneity), with objective response rate (ORR) at 12 weeks as defined via Response evaluation criteria in solid tumors (RECIST) 1.1 to pembrolizumab in patients with Programmed Death (PD)-1 inhibitor-naïve unresectable, American Joint Committee on Cancer (AJCC) stage III or distant metastatic (stage IV) melanoma.

Secondary Objectives

Estimate ORR (CR + PR) by RECIST 1.1 at 12 weeks to pembrolizumab in patients with PD-1 inhibitor-naïve unresectable stage III or distant metastatic metastatic melanoma (AJCC stage III/IV).

Estimate progression-free survival (PFS) in patients with unresectable stage III or distant metastatic melanoma treated with pembrolizumab as front-line therapy.

Explore associations in SUVmax and other PET parameters (e.g. total tumor metabolic volume, measurement of intra-tumoral and inter-lesional heterogeneity) between C11-AMT PET and fluorodeoxyglucose (FDG)-PET at baseline.

Explore associations between SUVmax, and other PET parameters (e.g. total tumor metabolic volume, measurement of intra-tumoral and inter-lesional heterogeneity) identified at baseline C11-AMT PET imaging with expression of components of the Indoleamine-pyrrole 2,3-dioxygenase (IDO) pathway detected by immunohistochemistry (IHC) or immunofluorescence (L -type amino acid transporter 1 (LAT1), IDO, tryptophan hydroxylase (TPH1)) and lymphocyte subtypes (CD4, cluster of differentiation 8 (CD8), FoxP3, MDSC), PD-1/PD-L1, and other immune checkpoint pathways (lymphocyte-associated gene 3 (LAG3), glucocorticoid-induced tumor necrosis factor receptor (GITR), T-cell immunoglobulin and mucin domain-3 (TIM3)) in freshly acquired tumor specimens prior to treatment with pembrolizumab.

Assess metabolic changes at week 12 (or earlier, if patient progresses) following treatment with pembrolizumab using baseline and week 12 FDG PET.

Outline:

Screening:

Physical exam, medical history, and laboratory tests, as per standard of care. Brain Magnetic resonance imaging (MRI) and Whole body FDG PET/ Computed tomography (CT) scan with IV contrast will be performed at least 24 hours before C11-AMT PET scanning. Although, the FDG PET/CT scan with IV contrast is preferred the following baseline measurements may be used if they have occurred within the below specified windows:

1. Whole body FDG PET/CT scan without IV contrast, will be accepted for study purposes (i.e. correlation between baseline FDG PET scan and baseline C11-AMT scan) if it has occurred within 28 days before the C11-AMT PET scan. In this case, the patient will only be required to have a baseline CT scan of the chest, abdomen, and pelvis (also neck, if applicable) with IV contrast within 28 days of starting pembrolizumab.
2. CT scan with intravenous (IV) contrast will be accepted for study purposes (i.e. baseline tumor assessment) if it has occurred within 28 days of starting pembrolizumab. In this case, the patient will only be required to have a baseline PET scan without CT coregistration 28 days prior to C11-AMT. This is to correlate baseline FDG PET with baseline C11-AMT PET parameters.

If eligibility criteria are met, patients will proceed to Study Related Scans and Biopsy:

C11-AMT PET will be performed at least 24 hours before pembrolizumab treatment and at least 24 hours after FDG PET/CT scan. A research biopsy will be performed before pembrolizumab treatment.

After screening and study related scans and biopsy, treatment will consist of the following:

Pembrolizumab 200mg IV flat dose will be administered over 30 minutes on Day 1; Pembrolizumab dosing will be repeated every 3 weeks until progression or subject withdrawal for other reasons.

At the end of treatment:

Whole body FDG PET/CT scan with IV contrast.

Projected Accrual:

Up to 25 subjects who have not received prior therapy for their recent diagnosis of distant metastatic melanoma.

ELIGIBILITY:
Inclusion Criteria:

1. Sign written informed consent and HIPAA authorization for release of personal health information. Note: HIPAA authorization may be included in the informed consent or obtained separately.
2. Subject must be 18 years of age or more on the day of signing informed consent.
3. Have histologic or cytologic biopsy-proven diagnosis of unresectable stage III or distant metastatic melanoma, irrespective of histologic type (i.e. cutaneous, unknown primary, mucosal, or ocular). Patients with resectable bulky stage IIIB or stage IIIC melanoma (for example at least 2.5-cm in shortest diameter for lymph nodes infiltrated by tumor and at least 2-cm in longest diameter for non-lymph nodes infiltrated by tumor) can also be entered into the study at the discretion of the Principal Investigator.
4. Have measurable disease based on RECIST v1.1. for solid tumors
5. Be willing to undergo fresh tumor tissue biopsy of an accessible tumor lesion prior to pembrolizumab. A mandatory fresh biopsy will be collected following C11-AMT PET imaging. Subjects for whom fresh samples cannot be provided (e.g. inaccessible or subject safety concern) or do not agree to this fresh tumor research biopsy of accessible tumor will be deemed ineligible for study participation. Exception to the mandatory tumor tissue collection are patients with metastatic lung lesions as the only site of metastatic disease. Fresh biopsy collection from these subjects will be optional, due to high risk of pneumothorax.
6. Be willing to allow for investigators to collect archival tumor tissues from surgical procedures that may have been performed before or after enrollment into this trial for research purposes (in-house cases and/or outside cases). These samples will be obtained by study staff as long as subject continues on follow-up. Blocks of tissue will be requested, and if blocks are not able to be obtained, 5micron slides (10-15) will be sufficient.
7. Be willing to be injected with 11C-methyl-L-tryptophan (C11-AMT)
8. Have a performance status of 0 - 2 on the Eastern Cooperative Oncology Group (ECOG) Performance Scale.
9. Has not received prior therapy with cytotoxic T lymphocyte antigen (CTLA)-4, PD-1/PD-L1 inhibitors, other co-stimulatory or co-inhibitory immune checkpoint antibody therapies (e.g. LAG3, TIM3, cluster of differentiation (CD) 137, Killer immunoglobulin-like receptor (KIR3DL), cluster of differentiation (CD) 70, and CD27) for distant metastatic melanoma. Patients who have received mitogen-activated protein kinase (MAPK) inhibitors are allowed on condition that they have recovered from adverse events to at most Grade 1 by CTCAE v4.03 and at least 15 days have elapsed between last dose of MAPK inhibitors and C11-AMT imaging. Patients who have previously received CTLA-4 inhibitors in the adjuvant setting are allowed to participate as long as they discontinued CTLA-4 treatment at least 30 days ago and meet criteria outlined in inclusion #14. Patients who have previously received adjuvant PD-1 inhibitors are excluded.
10. Demonstrate adequate organ function as defined in below; all screening labs to be obtained within 14 days prior to C11-AMT PET scan:

    Hematological:

    Hemoglobin (Hgb) - ≥ 9 g/dL or ≥ 5.6 mmol/L without transfusion or erythropoietin (EPO) dependency (within 7 days of Hgb) Absolute Neutrophil Count (ANC) - ≥ 1,500/mm3 Platelets - ≥ 100,000/mm3

    Renal:

    Serum Creatinine OR Measured or calculated creatinine clearance (GFR can also be used in place of creatinine or CrCl) - ≤1.5 x ULN OR ≥ 60 mL/min using the Cockcroft-Gault formula for subject with creatinine levels > 1.5 X institutional upper limits of normal (ULN)

    Hepatic:

    Serum Total Bilirubin - ≤ 1.5 X ULN Aspartate aminotransferase (AST) - ≤ 2.5 X ULN OR < 5 X ULN for subjects with liver metastases Alanine aminotransferase (ALT) - ≤ 2.5 X ULN OR < 5 X ULN for subjects with liver metastases Albumin - ≥ 2.5 mg/dL

    Coagulation:

    International Normalized Ratio (INR) or Prothrombin Time (PT) - ≤1.5 X ULN, unless subject is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants Activated Partial Thromboplastin Time (aPTT) - ≤1.5 X ULN, unless subject is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants
11. Female subjects of childbearing potential should have a negative urine or serum pregnancy within 14 days prior to C11-AMT PET scan. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
12. Female subjects of childbearing potential must be willing to use adequate methods of contraception as outlined - Contraception for the course of the study through 120 days after the last dose of study medication. Subjects of childbearing potential are those who have not been surgically sterilized or have not been free from menses for > 1 year.

    Note: Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the subject.

    Male subjects should agree to use an adequate method of contraception as outlined - Contraception starting with the first dose of study therapy through 120 days after the last dose of study therapy.

    Note: Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the subject.
13. Patients who have received prior adjuvant high dose interferon are allowed to participate as long as the last injection was given at least 30 days prior to the C11-AMT PET scan and they have fully recovered from side effects (i.e., Grade ≤1 or permanent side effects that require hormone replacement therapy).
14. Patients on adjuvant ipilimumab are allowed to participate at least 30 days from drug discontinuation as long as they have at most Grade 1 adverse events (or grade 2 if they have to received hormone replacement therapy for their otherwise grade 1 ipilimumab-induced autoimmune endocrinopathies).

Exclusion Criteria:

1. Is currently participating and receiving study therapy for his/her advanced melanoma or has participated in a study of an investigational agent and received study therapy in the advanced melanoma setting.
2. Has received prior treatment with PD-1/PD-L1 pathway inhibitors in the adjuvant setting.
3. Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to C11-AMT PET Scan
4. Has a known history of active tuberculosis (Bacillus Tuberculosis)
5. Hypersensitivity to pembrolizumab or any of its excipients described
6. Has had prior monoclonal antibody (mAb) targeting immune checkpoint proteins, for distant metastatic melanoma and have progressed or have developed intolerable side effect.
7. Adjuvant anticancer treatments are allowed at least 30 days has elapsed between the infusion/injection and C11-AMT PET scan as part of this study.
8. Prior radiation therapy for metastatic melanoma is allowed as long as the patient bears measurable actively growing disease outside the previously irradiated field. Note: If subject received major surgery, they must have recovered adequately from the toxicity (i.e., all symptoms ≤ grade 1) and/or complications from the intervention prior to starting therapy.
9. History of prior malignancy, with the exception of the following:

   * Non-melanoma skin cancers, non-invasive bladder cancer, and carcinoma in situ of the cervix,
   * Prior history of prostate provided patient not under active systemic treatment other than hormonal therapy and with documented undetectable prostate-specific antigen (PSA) (<0.2ng/mL),
   * Chronic lymphocytic leukemia (CLL)/ small lymphocytic lymphoma (SLL) provided patient has isolated lymphocytosis (Rai stage 0), and does not require systemic treatment [for "B" symptoms, Richter's transformation, lymphocyte doubling time (<6 months), lymphadenopathy or hepatosplenomegaly],
   * Lymphoma or any type or hairy-cell leukemia provided patient is not on active systemic treatment and is in complete remission, as evidenced by PET/CT scans and bone marrow biopsies for at least 3 months,
   * Papillary thyroid cancer. Since this malignancy very infrequently metastasizes distantly, patients with concurrent metastatic melanoma can be enrolled even if patients may: A) have just completed thyroidectomy within the last 2 years, B) have not received adjuvant radioactive iodine therapy, C) were only recently diagnosed with asymptomatic papillary thyroid cancer and their surgery is pending.
   * History of malignancy provided patient has completed therapy and is free of disease for ≥ 2 years. If patient had other malignancy within the last 2 years from which he may have been completely cured by surgery alone, he may considered to be enrolled on condition that the risk of development of distant metastatic disease based on AJCC staging system is less than 30%.
10. Has known active parenchymal central nervous system (CNS) metastases that are symptomatic, and/or more than one lesions, and/or their largest diameter is > 5-mm and/or require antiepileptic drugs or corticosteroids. Patients with carcinomatous meningitis are also excluded. Exceptions are: subjects with previously treated brain metastases provided they are stable (without evidence of progression by imaging) for at least 2 weeks prior to C11-AMT and any neurologic symptoms have returned to baseline, have no evidence of new or enlarging brain metastases, and are not using ongoing steroids for at least 7 days prior to C11-AMT. Patients with active (i.e. not treated with stereotactive radiosurgery), single, asymptomatic, up to 5-mm in largest diameter brain metastases (measured either by brain MRI with IV contrast or head CT with IV contrast measured within 2 weeks prior to C11-AMT) are allowed.
11. Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease-modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
12. Has known history of (non-infectious) pneumonitis that required steroids, or any evidence of current pneumonitis.
13. Has an active infection requiring systemic therapy.
14. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
15. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
16. Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment.
17. Has a known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies).
18. Has known active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C virus (HCV) (e.g., HCV RNA [qualitative] is detected).
19. Has received a live vaccine within 14 days of C11-AMT PET scan. Note: Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however intranasal influenza vaccines (e.g., Flu-Mist®) are live attenuated vaccines, and are not allowed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2017-04-19 (Actual); Primary Completion 2021-04-01 (Actual); Study Completion 2023-07-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stergios Moschos, MD, Principal Investigator — Department of Medicine, Division of Hematology/Oncology, University of North Carolina at Chapel Hill
Locations (2):
- United States (2):
  - Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - UNC Rex Healthcare, Raleigh, North Carolina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Oldan JD, Giglio BC, Smith E, Zhao W, Bouchard DM, Ivanovic M, Lee YZ, Collichio FA, Meyers MO, Wallack DE, Abernethy-Leinwand A, Long PK, Trembath DG, Googe PB, Kowalski MH, Ivanova A, Ezzell JA, Nikolaishvili-Feinberg N, Thomas NE, Wong TZ, Ollila DW, Li Z, Moschos SJ. Increased tryptophan, but not increased glucose metabolism, predict resistance of pembrolizumab in stage III/IV melanoma. Oncoimmunology. 2023 Apr 26;12(1):2204753. doi: 10.1080/2162402X.2023.2204753. eCollection 2023. PMID 37123046
- See also: University of North Carolina Lineberger Comprehensive Cancer Center Clinical Trials — https://unclineberger.org/patientcare/clinical-trials

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from 5/31/2017 through 11/06/2020 at two cancer centers in North Carolina. Subjects were enrolled in the study between 06/01/2017 -11/11/2020.
Pre-assignment Details: A total of thirty-three participants consented to the study, but five were deemed to be ineligible and one withdrawn the consent during screening, and therefore were not enrolled on the study.
Period: Overall Study
Arm/Group | Single Arm
Started | 27
Completed | 26
Not Completed | 1
Not completed — Progression after Cycle 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Single Arm: This is a single-arm study. All participants completed all the study interventions namely pembrolizumab treatment, FDG PET, C11-AMT PET, and CT scans.
Arm/Group | Single Arm
Number analyzed (Participants) | 27
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 16
  >=65 years | 11
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 21
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 27
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 26
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 27

OUTCOME MEASURES:

1. Primary Outcome: Association of Baseline C11-AMT PET SUV Max Value With Objective Response
Description: Association between intensity of C11-AMT PET at baseline, as measured by maximum standardized uptake value (SUV max) and objective response (OR) using computerized tomography images with intravenous contrast, as defined via RECIST v.1.1, at 12 weeks. Subject is considered responder if subject has CR or PR while subject is considered not-responder if they do not have CR or PR at 12 weeks.
  RECIST v.1.1: Complete Response (CR), disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Stable Disease (SD), no response or less response than Partial or Progressive; or Progressive Disease (PD), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: 12 weeks
Population: Participants who received study treatment and pretreatment C11-AMT PET scanning performed, and tumor response assessed according to RECIST v1.1. criteria based on the CT scan with IV contrast, 12 weeks after starting treatment.
  C11-AMT PET SUV max cut-off value = 5 was selected considering optimal cut-point analysis, based on whether participants remained free of recurrence while on study treatment or lived longer, demonstrated "higher" or "lower" C11-AMT SUV max.
Measure: Count of Participants; unit: Participants
Groups:
- Baseline C11AMT PET SUVmax<5: Baseline 11C-methyl-L-tryptophan (C11-AMT) positron emission tomography (PET) maximum standardized uptake value (SUVmax) is less than 5.
- Baseline C11AMT PET SUVmax>5: Baseline 11C-methyl-L-tryptophan (C11-AMT) positron emission tomography (PET) maximum standardized uptake value (SUVmax) is bigger than 5.
Arm/Group | Baseline C11AMT PET SUVmax<5 | Baseline C11AMT PET SUVmax>5
Number analyzed (Participants) | 7 | 19
Participants
  Responder | 6 | 6
  Not-Responder | 1 | 13
Statistical Analysis 1: Comparison: Baseline C11AMT PET SUVmax<5 vs Baseline C11AMT PET SUVmax>5; Null hypothesis. No association between baseline C11-AMT PET SUVmax value and antitumor response to pembrolizumab; Test type: Other — 2-tailed Fisher's exact test; p = 0.08, 2-tailed Fisher's exact test

2. Secondary Outcome: Objective Response Rate
Description: Objective Response Rate (ORR) is defined as the number of the subjects with a Complete Response, Partial Response, stable disease, and progressive disease according to Response Evaluation Criteria in Solid Tumors ( RECIST 1.1) at 12 weeks after starting to study treatment.
  RECIST v.1.1: Complete Response (CR), disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Stable Disease (SD), no response or less response than Partial or Progressive; or Progressive Disease (PD), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: 12 Weeks
Population: Subjects received at least one dose of the study treatment and response evaluation according to RECIST 1.1 at 12 weeks, were performed.
Measure: Count of Participants; unit: Participants
Arm/Group | Single Arm
Number analyzed (Participants) | 26
Participants
  Complete response | 7
  Partial response | 5
  Stable Disease | 2
  Progressive Disease | 12

3. Secondary Outcome: Progression-Free Survival
Description: Progression Free Sruvival (PFS) is defined time from first day of treatment until disease progression as defined by RECIST1.1.
Time Frame: 3 years
Population: The subjects received at least one dose of the study treatment and treatments response was assessed.
Measure: Median (Full Range); unit: months
Arm/Group | Single Arm
Number analyzed (Participants) | 26
months | 7.4 [0.6 to 52.6]

4. Secondary Outcome: Association of Baseline FDG-PET and C11-AMT PET
Description: Associations of SUVmax values between baseline FDG-PET and baseline C11-AMT PET images were examined.
  To objectively determine tumor regions of interest on C11-AMT and 18F FDG PET, the voxel with the highest tracer concentration (e.g., SUVmax) was determined. The voxel with the highest AMT tracer concentration (e.g., SUVmax) as well as a background region in close proximity to the location of the tumor using the MIM vista PET viewing software (MIM software Inc., Cleveland, OH, version 7.0.5).
Time Frame: Baseline
Population: All the tumor lesions with measured/determined SUVmax values belong to subjects who underwent baseline C11 AMT PET and FDG PET images were included.
Measure: Median (Full Range); unit: units on a scale
Units Other Than Participants: Total number of tumor lesions analyzed
Groups:
- FDG PET SUVmax: Baseline FDG PET SUVmax (ratio above background)
- C11AMT PET SUVmax: Baseline C11AMT PET SUVmax (ratio above background)
Arm/Group | FDG PET SUVmax | C11AMT PET SUVmax
Number analyzed (Participants) | 26 | 26
Number analyzed (Total number of tumor lesions analyzed) | 61 | 61
units on a scale | 8.5 [2.1 to 28] | 5.3 [3.1 to 23]

5. Secondary Outcome: Metabolic Changes
Description: Assess metabolic changes at week 12 (or earlier, if patient progresses) following treatment with pembrolizumab using baseline and week 12 FDG PET. Each lesion is considered independently since subjects might have some lesion with SUV max value increased and another lesion with SUV max value decreased.
Time Frame: 12 weeks
Population: Tumor lesions from the subjects who participated in the trial had available FDG PET data before and after 12 weeks ofpembrolizumab treatment (or earlier, if progression). Fifty-two tumor lesions from 23 subjects were analyzed.
Measure: Count of Units; unit: Number of tumor lesions
Units Other Than Participants: Number of tumor lesions
Groups:
- SUVmax Increased: Baseline FDG PET SUVmax valueincreased, at week 12.
- SUVmax Decreased: Baseline FDG PET SUVmax valuedecreased, at week 12.
Arm/Group | SUVmax Increased | SUVmax Decreased
Number analyzed (Participants) | 23 | 23
Number analyzed (Number of tumor lesions) | 20 | 32
Number of tumor lesions
  Responder | 1 | 30
  Stable | 1 | 0
  Not-Responder | 18 | 2

6. Secondary Outcome: Baseline Positron Emission Tomography (PET) Parameters (SUVmax) Corresponding to Tumors That Were Subsequently Collected for Immunohistochemical (IHC) Analysis. Melanoma-specific Indoleamine 2,3-dioxygenase (IDO) Protein Expression in Research Biopsies
Description: Outcome Measure Description: Associations between baseline C-methyl-L-tryptophan (C11-AMT) PET imaging and fluorodeoxyglucose (FDG) PET SUVmax values with melanoma-specific IDO expression by single colon immunohistochemistry (IHC) within the harvested tumors.
  We used the following single-color IHC scoring system to semiquantify the staining intensity and percentage of positive melanoma cells: 0 (no staining), 1+ (<25% of melanoma cells with membrane or cytoplasmic stain), 2+ (25-80% of melanoma cells with the membrane of cytoplasmic stain), 3+ (>80% of melanoma cells with membrane or cytoplasmic stain) scale was used.
Time Frame: Baseline
Population: Research tumor specimens that were collected from patients who enrolled into the study, had been previously imaged with C11-AMT PET and FDG PET imaging, and were available/suitable for IHC analysis for IDO expression by IHC. Of the 26 tumor specimens, only 18 had sufficient tumor for correlation analysis.
Measure: Median (Full Range); unit: score on a scale
Groups:
- Baseline FDG PET SUVmax: The baseline FDG SUVmax value and the single-color IDO IHC staining score
- C11-AMT SUVmax: The baseline C11-AMT SUVmax value and the single-color indoleamine 2,3-dioxygenase pathway immunohistochemistry staining score.
Arm/Group | Baseline FDG PET SUVmax | C11-AMT SUVmax
Number analyzed (Participants) | 18 | 18
score on a scale
  IDO score 0: number analyzed (Participants) | 5 | 5
  IDO score 0 | 9.8 [2.7 to 20] | 5.9 [4.1 to 23]
  IDO score 1: number analyzed (Participants) | 8 | 8
  IDO score 1 | 8.65 [4.3 to 19] | 7.8 [3.6 to 21]
  IDO score 2: number analyzed (Participants) | 4 | 4
  IDO score 2 | 7.35 [5.7 to 21.8] | 3.7 [3.3 to 12.9]
  IDO score 3: number analyzed (Participants) | 1 | 1
  IDO score 3 | 3.4 [3.4 to 3.4] | 3.1 [3.1 to 3.1]

ADVERSE EVENTS:
Time Frame: Up to 114 days.
Description: Adverse events were collected from day one of the study drug administration to 30 days after completion of treatment.
Arm/Group | Single Arm
All-Cause Mortality (participants affected / at risk) | 9/27
Serious Adverse Events (participants affected / at risk) | 5/27
Other Adverse Events (participants affected / at risk) | 27/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Single Arm (N=27)
Neoplasms benign, malignant and unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1
Neutrophil count decreased (Investigations) | 1
Retinal detachment (Eye disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Single Arm (N=27)
Anemia (Blood and lymphatic system disorders) | 5
Cardiac disorders - Other, specify (Cardiac disorders) | 1
Chest pain - cardiac (Cardiac disorders) | 1
Hearing impaired (Ear and labyrinth disorders) | 1
Vertigo (Ear and labyrinth disorders) | 2
Endocrine disorders - Other, specify (Endocrine disorders) | 1
Hyperthyroidism (Endocrine disorders) | 4
Hypothyroidism (Endocrine disorders) | 2
Blurred vision (Eye disorders) | 3
Eye disorders - Other, specify (Eye disorders) | 1
Floaters (Eye disorders) | 1
Retinal detachment (Eye disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 3
Constipation (Gastrointestinal disorders) | 5
Diarrhea (Gastrointestinal disorders) | 5
Dry mouth (Gastrointestinal disorders) | 1
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 5
Vomiting (Gastrointestinal disorders) | 1
Edema limbs (General disorders) | 3
Facial pain (General disorders) | 2
Fatigue (General disorders) | 24
Flu like symptoms (General disorders) | 1
Localized edema (General disorders) | 2
Pain (General disorders) | 11
Hepatic pain (Hepatobiliary disorders) | 1
Immune system disorders - Other, specify (Immune system disorders) | 1
Infections and infestations - Other, specify (Infections and infestations) | 2
Papulopustular rash (Infections and infestations) | 1
Seroma (Injury, poisoning and procedural complications) | 1
Alanine aminotransferase increased (Investigations) | 5
Alkaline phosphatase increased (Investigations) | 1
Aspartate aminotransferase increased (Investigations) | 6
Blood bilirubin increased (Investigations) | 4
Creatinine increased (Investigations) | 2
Investigations - Other, specify (Investigations) | 3
Lymphocyte count decreased (Investigations) | 13
Neutrophil count decreased (Investigations) | 2
Platelet count decreased (Investigations) | 1
White blood cell decreased (Investigations) | 5
Anorexia (Metabolism and nutrition disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 2
Hypercalcemia (Metabolism and nutrition disorders) | 2
Hyperglycemia (Metabolism and nutrition disorders) | 2
Hyperkalemia (Metabolism and nutrition disorders) | 4
Hypertriglyceridemia (Metabolism and nutrition disorders) | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 1
Hyponatremia (Metabolism and nutrition disorders) | 2
Metabolism and nutrition disorders - Other, specify (Metabolism and nutrition disorders) | 2
Obesity (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 4
Arthritis (Musculoskeletal and connective tissue disorders) | 3
Back pain (Musculoskeletal and connective tissue disorders) | 2
Bone pain (Musculoskeletal and connective tissue disorders) | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 2
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 4
Neck pain (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Dizziness (Nervous system disorders) | 4
Dysesthesia (Nervous system disorders) | 1
Dysgeusia (Nervous system disorders) | 1
Headache (Nervous system disorders) | 6
Ischemia cerebrovascular (Nervous system disorders) | 1
Paresthesia (Nervous system disorders) | 1
Peripheral sensory neuropathy (Nervous system disorders) | 1
Anxiety (Psychiatric disorders) | 4
Depression (Psychiatric disorders) | 1
Insomnia (Psychiatric disorders) | 3
Psychiatric disorders - Other, specify (Psychiatric disorders) | 1
Chronic kidney disease (Renal and urinary disorders) | 1
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 1
Urinary frequency (Renal and urinary disorders) | 2
Reproductive system and breast disorders - Other, specify (Reproductive system and breast disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 1
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 1
Sleep apnea (Respiratory, thoracic and mediastinal disorders) | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1
Dry skin (Skin and subcutaneous tissue disorders) | 3
Pruritus (Skin and subcutaneous tissue disorders) | 11
Rash acneiform (Skin and subcutaneous tissue disorders) | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 7
Scalp pain (Skin and subcutaneous tissue disorders) | 1
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 5
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 2
Surgical and medical procedures - Other, specify (Surgical and medical procedures) | 2
Hot flashes (Vascular disorders) | 2
Hypertension (Vascular disorders) | 5
Lymphedema (Vascular disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-03-12): https://cdn.clinicaltrials.gov/large-docs/06/NCT03089606/Prot_SAP_000.pdf